CLINICAL TRIAL: NCT07282782
Title: A Prospective, Randomized Parallel Group Study of the Efficacy of Vancomycin Administered Through Intraarticular Injection Versus Intraosseous Injection Versus Intravenous Infusion in Patients Undergoing Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Scott Ball, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 810594
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-10

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intravenous (IV) Vancomycin (No Intervention): Standard of care dose based on patient weight, organ function, and clinical factors at the discretion of the treating physician
- Intraosseous (IO) Vancomycin (Experimental): 500mg dose Vancomycin (in 100mL saline)
  Interventions: Drug: Vancomycin
- Intraarticular (IA) Vancomycin (Experimental): 500mg dose Vancomycin (in 30mL saline)
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — Intraosseous or Intraarticular administration of Vancomycin
  Arms: Intraarticular (IA) Vancomycin; Intraosseous (IO) Vancomycin

SUMMARY:
Periprosthetic joint infection (PJI) is a national health crisis and leads to very poor outcomes for patients undergoing elective joint replacement. Within the realm of elective total knee arthroplasty (TKA), various methods of infection prophylaxis are in place. These include sterile precautions, would/tissue handling, and antibiotic prophylaxis. With respect to the latter, various approaches have been utilized including intravenous and intraosseous administration of vancomycin, preoperatively. Intraosseous administration does require another wound and a specific device to administer. We proposed that intraarticular injection of vancomycin is non-inferior to intraosseous administration, thus reducing wounds, time, and cost.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 years of age receiving treatment at UC San Diego Health
* Undergoing primary unilateral TKA
* Ability to provide consent

Exclusion Criteria:

* previous surgery on the knee (with the exception of arthroscopy)
* BMI > 35
* contraindication to receiving vancomycin, cefepime or cefazolin (ie, allergy, etc)
* diabetics with A1c>7.5% (unless controlled fructosamine)
* immunocompromised or immunosuppressed patients (HIV, Hepatitis C, end stage renal disease (ESRD), post transplant, chemotherapy or radiation therapy within 6 months of surgery, immunomodulating meducations)
* no history of active infections
* no history of chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of vancomycin in bone, synovial tissue, subcutaneous fat and serum blood | Intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States